CLINICAL TRIAL: NCT01442064
Title: An Open-Label, Multicenter Extension Study to Evaluate the Safety and Tolerability of Ranibizumab in Subjects With Choroidal Neovascularization (CNV) Secondary to Age-Related Macular Degeneration (AMD) or Macular Edema Secondary to Retinal Vein Occlusion (RVO) Who Have Completed a Genentech-Sponsored Ranibizumab Study
Brief Title: An Extension Study to Evaluate Safety and Tolerability of Ranibizumab in Macular Edema Secondary to Retinal Vein Occlusion (Cohort 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF3426g (Cohort 2)
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Results first posted 2012-01-10 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2011-12

CONDITIONS: Macular Edema; Retinal Vein Occlusion
Keywords: CNV; Lucentis; AMD; Age-related macular degeneration; RVO; Macular edema secondary to retinal vein occlusion
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion; Macular Degeneration | interventions — Ranibizumab

ARMS (1):
- Ranibizumab 0.5 mg (Experimental): Ranibizumab 0.5 mg intravitreal injection administered as-needed no more frequently than every 30 days (no more than 12 injections per year) for 24 months.
  Interventions: Drug: Ranibizumab 0.5 mg

INTERVENTIONS:
Drug: Ranibizumab 0.5 mg — Ranibizumab intravitreal injection 0.5 mg in a single-dose regimen given on an as needed basis no more frequently than every 30 days (no more than 12 injections per year).
  Other Names: Lucentis

SUMMARY:
This is an open-label, multicenter, extension study of intravitreally administered ranibizumab in two cohorts. The first cohort (reported separately under FVF3426g, NCT00379795) enrolled subjects with primary or recurrent Choroidal Neovascularization (CNV) secondary to Age-Related Macular Degeneration (AMD) who completed the treatment phase of a Genentech sponsored study (FVF2598g (NCT00056836), FVF2587g (NCT00061594), or FVF2428g (NCT00056823)). The second cohort (reported here) enrolled subjects with macular edema secondary to Retinal Vein Occlusion (RVO) who completed the 6-month treatment and 6-month observation phases (12 months total) of a Genentech sponsored study (FVF4165g (NCT00486018) or FVF4166g (NCT00485836)). Patients were enrolled within 14 days of completion of the previous study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* The 6-month treatment and 6-month observation phases (12 months total) of a Genentech-sponsored ranibizumab study for RVO (FVF4165g or FVF4166g)
* Expectation by the investigator that the subject may potentially benefit from intravitreal anti-vascular endothelial growth factor (VEGF) treatment

Exclusion Criteria:

* History of intraocular surgery (including cataract extraction, scleral buckle, etc.) within 1 month prior to Day 0 of this extension study
* Concurrent use of systemic anti-VEGF agents
* Use of RVO treatments not approved by the Food and Drug Administration (FDA) in the study eye
* Use of intravitreal bevacizumab in the study eye and/or fellow eye
* Macular edema in the study eye due to other causes than RVO such as diabetes
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 30 mmHg despite treatment with antiglaucoma medication)
* Pregnancy or lactation
* Premenopausal women not using adequate contraception
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications
* Current treatment for active systemic infection
* Inability to comply with study or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Lai, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an open label multi-center extension study for participants who completed FVF4165g BRAVO (NCT00486018) or FVF4166g CRUISE (NCT0048583). Cohort 2 consists of enrolled participants with macular edema secondary to retinal vein occlusion (RVO).
Groups:
- Ranibizumab (Sham BRAVO): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as-needed no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received intravitreal sham injections in the 6 month treatment period of BRAVO and received ranibizumab in the 6 month observation period of BRAVO or in this extension study.
- Ranibizumab (0.3 mg BRAVO): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as-needed no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received 0.3 mg Ranibizumab intravitreal injections in the 6 month treatment period of BRAVO.
- Ranibizumab (0.5 mg BRAVO): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as-needed no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received 0.5 mg Ranibizumab intravitreal injections in the 6 month treatment period of BRAVO.
- Ranibizumab (Sham CRUISE): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as-needed no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received intravitreal sham injections in the 6 month treatment period of CRUISE and received ranibizumab in the 6 month observation period of CRUISE or in this extension study.
- Ranibizumab (0.3 mg CRUISE): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as-needed no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received 0.3 mg Ranibizumab intravitreal injections in the 6 month treatment period of CRUISE.
- Ranibizumab (0.5 mg CRUISE): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as-needed no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received 0.5 mg Ranibizumab intravitreal injections in the 6 month treatment period of CRUISE.
Period: Overall Study
Arm/Group | Ranibizumab (Sham BRAVO) | Ranibizumab (0.3 mg BRAVO) | Ranibizumab (0.5 mg BRAVO) | Ranibizumab (Sham CRUISE) | Ranibizumab (0.3 mg CRUISE) | Ranibizumab (0.5 mg CRUISE)
Started | 97 | 103 | 104 | 98 | 107 | 99
Ranibizumab-Treated Subjects | 93 (Includes participants who received Ranibizumab in either the initial studies or the extension study.) | 103 | 104 | 96 | 107 | 99
Received Study Drug in Extension Study | 61 | 70 | 60 | 70 | 89 | 81
Completed | 0 | 2 | 0 | 0 | 1 | 0
Not Completed | 97 | 101 | 104 | 98 | 106 | 99
Not completed — Adverse Event | 2 | 2 | 2 | 1 | 2 | 0
Not completed — Death | 0 | 1 | 3 | 3 | 1 | 3
Not completed — Lost to Follow-up | 5 | 5 | 1 | 1 | 3 | 3
Not completed — Physician Decision | 1 | 1 | 2 | 3 | 3 | 1
Not completed — Withdrawal by Subject | 6 | 3 | 2 | 2 | 2 | 1
Not completed — Sponsor decision | 82 | 88 | 92 | 88 | 95 | 87
Not completed — Subject non-compliance | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Condition mandated other intervention | 1 | 1 | 2 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Ranibizumab (Sham BRAVO): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as needed no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received intravitreal sham injections in the 6 month treatment period of BRAVO and received ranibizumab in the 6 month observation period of BRAVO or in this extension study.
- Ranibizumab (0.3 mg BRAVO): In this extension study participant received Ranibizumab 0.5 mg intravitreal injection administered as needed no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received 0.3 mg Ranibizumab intravitreal injections in the 6 month treatment period of BRAVO.
- Ranibizumab (0.5 mg BRAVO): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as needed no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received 0.5 mg Ranibizumab intravitreal injections in the 6 month treatment period of BRAVO.
- Ranibizumab (Sham CRUISE): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as needed no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received intravitreal sham injections in the 6 month treatment period of CRUISE and received ranibizumab in the 6 month observation period of CRUISE or in this extension study.
- Total: Total of all reporting groups
Arm/Group | Ranibizumab (Sham BRAVO) | Ranibizumab (0.3 mg BRAVO) | Ranibizumab (0.5 mg BRAVO) | Ranibizumab (Sham CRUISE) | Ranibizumab (0.3 mg CRUISE) | Ranibizumab (0.5 mg CRUISE) | Total
Number analyzed (Participants) | 97 | 103 | 104 | 98 | 107 | 99 | 608
Age, Customized [Number; unit: participants]
  <45 years | 5 | 3 | 3 | 8 | 3 | 4 | 26
  45 to <65 years | 43 | 39 | 38 | 37 | 26 | 32 | 215
  65 to <85 years | 45 | 54 | 55 | 49 | 68 | 59 | 330
  ≥85 years | 4 | 7 | 8 | 4 | 10 | 4 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 57 | 46 | 41 | 52 | 39 | 278
  Male | 54 | 46 | 58 | 57 | 55 | 60 | 330

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ocular Adverse Events in the Study Eye
Description: Number of participants with: any ocular adverse events, ocular adverse events causing treatment discontinuation, ocular serious adverse events, intraocular inflammation and cataracts that occurred in the study eye.
  Only adverse events that occurred during this extension study are reported. For subjects in the crossover groups who started their first ranibizumab injection in this extension study, adverse events that occurred prior to any ranibizumab injection were also excluded.
Time Frame: Up to 24 months
Population: Ranibizumab- Treated Participants includes all participants who received Ranibizumab in one of the initial studies or this extension study. This analysis includes only those adverse events that occurred during this extension study.
Measure: Number; unit: participants
Groups:
- Ranibizumab (0.3 mg BRAVO): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection as-needed administered no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received 0.3 mg Ranibizumab intravitreal injections in the 6 month treatment period of BRAVO.
- Ranibizumab (0.5 mg BRAVO): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection as-needed administered no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received 0.5 mg Ranibizumab intravitreal injections in the 6 month treatment period of BRAVO.
- Ranibizumab (Sham CRUISE): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as-needed no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received sham intravitreal injections in the 6 month treatment period of CRUISE and received ranibizumab in the 6 month observation period of CRUISE or in this extension study.
- Ranibizumab (0.5 mg CRUISE): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection as-needed administered no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received 0.5 mg Ranibuzumab intravitreal injections in the 6 month treatment period of CRUISE.
Arm/Group | Ranibizumab (Sham BRAVO) | Ranibizumab (0.3 mg BRAVO) | Ranibizumab (0.5 mg BRAVO) | Ranibizumab (Sham CRUISE) | Ranibizumab (0.3 mg CRUISE) | Ranibizumab (0.5 mg CRUISE)
Number analyzed (Participants) | 93 | 103 | 104 | 96 | 107 | 99
participants
  Any ocular adverse event (AE) | 51 | 64 | 63 | 60 | 67 | 66
  Ocular AE leading to treatment discontinuation | 1 | 2 | 2 | 0 | 2 | 2
  Ocular serious adverse event | 2 | 4 | 6 | 5 | 10 | 3
  Intraocular inflammation | 0 | 0 | 0 | 2 | 3 | 1
  Cataract | 6 | 10 | 6 | 3 | 6 | 5

2. Primary Outcome: Number of Participants With Non-ocular Adverse Events
Description: Number of participants with non-ocular adverse events (not occurring in the eye) in the following categories: any adverse events, serious adverse events, adverse events leading to study discontinuation and death.
  Only adverse events that occurred during this extension study are reported. For subjects in the crossover groups who started their first ranibizumab injection in this extension study, adverse events that occurred prior to any ranibizumab injection were also excluded.
  Additional information about adverse events can be found in the adverse events section.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ranibizumab (Sham BRAVO) | Ranibizumab (0.3 mg BRAVO) | Ranibizumab (0.5 mg BRAVO) | Ranibizumab (Sham CRUISE) | Ranibizumab (0.3 mg CRUISE) | Ranibizumab (0.5 mg CRUISE)
Number analyzed (Participants) | 93 | 103 | 104 | 96 | 107 | 99
participants
  Any non-ocular adverse event | 56 | 77 | 68 | 58 | 71 | 64
  Serious non-ocular adverse event | 10 | 15 | 18 | 16 | 21 | 20
  Non-ocular adverse event led to discontinuation | 1 | 0 | 1 | 0 | 1 | 0
  Death | 0 | 1 | 3 | 3 | 1 | 3

3. Secondary Outcome: Change From Baseline in the Best Corrected Visual Acuity (BCVA)
Description: Change from baseline in then BCVA was assessed by the number of letters a patient could read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) Eye Chart at a Starting Test Distance of 4 Meters. An increase in the number of letters read indicates improvement in visual acuity.
Time Frame: Baseline (Day 0 of extension study), Months 6, 12, 18, and 24
Population: Enrolled participants for whom data was available for analyses at the given time-points. Observed data were used with no imputation. The number of participants for whom data was available for analyses is represented by "n".
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab (Sham BRAVO) | Ranibizumab (0.3 mg BRAVO) | Ranibizumab (0.5 mg BRAVO) | Ranibizumab (Sham CRUISE) | Ranibizumab (0.3 mg CRUISE) | Ranibizumab (0.5 mg CRUISE)
Number analyzed (Participants) | 97 | 103 | 104 | 98 | 107 | 99
letters
  Month 6 (n=88,96,98,90,101,91) | -0.1 (8.1) | -2.2 (10.5) | -1.3 (7.1) | -3.2 (10.4) | -4.1 (10.7) | -3.2 (9.7)
  Month 12 (n=66,66,73,58,69,50) | 0.9 (6.9) | -2.3 (11.5) | -0.7 (7.3) | -4.2 (11.3) | -5.2 (13.8) | -4.1 (12.9)
  Month 18 (n=23,26,32,31,26,22) | 0.5 (5.0) | -1.7 (6.3) | -6.1 (15.5) | -5.1 (14.6) | -6.1 (12.1) | -0.8 (10.9)
  Month 24 (n=0,2,0,0,1,0) | NA (NA) — No participants with data available for this time point. | -4.5 (16.3) | NA (NA) — No participants with data available for this time point. | NA (NA) — No participants with data available for this time point. | -1.0 (NA) — Only 1 participant in this group. Standard deviation not calculated. | NA (NA) — No participants with data available for this time point.

4. Secondary Outcome: Change From Baseline in Central Foveal Thickness at Month 6 and Month 12
Description: Change from baseline in Central foveal (retinal) thickness was assessed by Optical Coherence Tomography (OCT). OCT was conducted at the study sites by personnel who were certified by the University of Wisconsin Fundus Photograph Reading Center.
Time Frame: Baseline (Day 0 of extension study), Months 6 and 12
Population: Enrolled participants for whom data was available for analyses at the given time-point as indicated by "n" in the categories. Observed data were used with no imputation.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Ranibizumab (Sham BRAVO) | Ranibizumab (0.3 mg BRAVO) | Ranibizumab (0.5 mg BRAVO) | Ranibizumab (Sham CRUISE) | Ranibizumab (0.3 mg CRUISE) | Ranibizumab (0.5 mg CRUISE)
Number analyzed (Participants) | 97 | 103 | 104 | 98 | 107 | 99
µm
  Month 6 (n=86,96,97,90,101,89) | 21.5 (131.6) | 36.8 (159.8) | 40.2 (117.4) | 87.4 (217.1) | 161.4 (289.1) | 94.6 (235.9)
  Month 12 (n=62,65,72,56,69,51) | 3.7 (124.9) | 6.3 (163.7) | 35.3 (110.6) | 79.7 (199.4) | 88.3 (262.9) | 68.4 (252.7)

5. Secondary Outcome: Change From Baseline in Visual Function Composite Score, as Measured by the National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25)
Description: NEI VFQ-25 is a 25 item questionnaire that assesses visual function and quality of life for a total possible score of 0 to 100. A higher score represents better functioning. The change from baseline is calculated at Month 12 and Month 24.
  Participants are grouped according to the treatment they received in initial studies FVF4165g BRAVO (NCT00486018) and FVF4166g CRUISE (NCT00485836).
Time Frame: Baseline (Day 0 of extension study), Months 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Ranibizumab (Sham BRAVO): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as-needed no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Participants in this group received intravitreal sham injections in the 6 month treatment period of BRAVO and received ranibizumab in the 6 month observation period of BRAVO or in this extension study.
- Ranibizumab (0.3 mg BRAVO): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection as-needed administered no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Participants in this group received 0.3 mg Ranibizumab intravitreal injections in the 6 month treatment period of BRAVO.
- Ranibizumab (0.5 mg BRAVO): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection as-needed administered no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Participants in this group received 0.5 mg Ranibizumab intravitreal injections in the 6 month treatment period of BRAVO.
- Ranibizumab (Sham CRUISE): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as-needed no more frequently than every 30 days (no more than 12 injections per year)for 24 months. Participants in this group received sham intravitreal injections in the 6 month treatment period of CRUISE and received ranibizumab in the 6 month observation period of CRUISE or in this extension study.
- Ranibizumab (0.3 mg CRUISE): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as-needed no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Participants in this group received 0.3 mg Ranibizumab intravitreal injections in the 6 month treatment period of CRUISE.
- Ranibizumab (0.5 mg CRUISE): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection as-needed administered no more frequently than every 30 days (no more than 12 injections per year) for 24 months. Participants in this group received 0.5 mg Ranibuzumab intravitreal injections in the 6 month treatment period of CRUISE.
Arm/Group | Ranibizumab (Sham BRAVO) | Ranibizumab (0.3 mg BRAVO) | Ranibizumab (0.5 mg BRAVO) | Ranibizumab (Sham CRUISE) | Ranibizumab (0.3 mg CRUISE) | Ranibizumab (0.5 mg CRUISE)
Number analyzed (Participants) | 97 | 103 | 104 | 98 | 107 | 99
Scores on a scale
  Month 12 (n=64,65,72,58,67,50) | -0.3 (10.0) | -0.7 (9.7) | -0.7 (8.6) | 0.1 (10.5) | -1.0 (8.0) | -1.6 (7.7)
  Month 24 (n=0,2,0,0,1,0) | NA (NA) — No participants with data available for this time point. | 6.2 (7.4) | NA (NA) — No participants with data available for this time point. | NA (NA) — No participants with data available for this time point. | -13.3 (NA) — Only 1 participant with data available in this group. Standard deviation not calculated. | NA (NA) — No participants with data available for this time point.

ADVERSE EVENTS:
Time Frame: Up to 24 months
Description: Safety Population included all participants who received at least one dose of study drug in one of the initial studies or this extension study. These analyses include only those adverse events that occurred during this extension study.
Groups:
- Ranibizumab (Sham): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as-needed no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received intravitreal sham injections in the 6 month treatment period of BRAVO or the 6 month treatment period of CRUISE and received Ranibizumab during the 6 month observation period of the initial study or this extension study.
- Ranibizumab (0.3 mg): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as-needed no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received 0.3 mg Ranibizumab intravitreal injections in the 6 month treatment period of BRAVO or the 6 month treatment period of CRUISE.
- Ranibizumab (0.5 mg): In this extension study participants received Ranibizumab 0.5 mg intravitreal injection administered as-needed no more frequently than every 30 days (no more than 12 injections per year) up to 24 months. Participants in this group received 0.5 mg Ranibizumab intravitreal injections in the 6 month treatment period of BRAVO or the 6 month treatment period of CRUISE.
Arm/Group | Ranibizumab (Sham) | Ranibizumab (0.3 mg) | Ranibizumab (0.5 mg)
Serious Adverse Events (participants affected / at risk) | 32/189 | 49/210 | 46/203
Other Adverse Events (participants affected / at risk) | 146/189 | 179/210 | 172/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (Sham) (N=189) | Ranibizumab (0.3 mg) (N=210) | Ranibizumab (0.5 mg) (N=203)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 2 | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 | 0 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 1 | 3
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 0 | 1
COR PULMONALE (Cardiac disorders) | 0 | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 2 | 0 | 2
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 1
SINUS ARRHYTHMIA (Cardiac disorders) | 1 | 0 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1
AMAUROSIS FUGAX (Eye disorders) | 0 | 1 | 0
CATARACT (Eye disorders) | 0 | 1 | 0
CYSTOID MACULAR OEDEMA (Eye disorders) | 0 | 1 | 0
MACULAR ISCHAEMIA (Eye disorders) | 0 | 1 | 0
MACULAR OEDEMA (Eye disorders) | 1 | 2 | 4
MACULOPATHY (Eye disorders) | 0 | 0 | 1
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 0 | 1 | 1
RETINAL VEIN OCCLUSION (Eye disorders) | 0 | 2 | 1
VISUAL ACUITY REDUCED (Eye disorders) | 4 | 3 | 2
VISUAL ACUITY REDUCED TRANSIENTLY (Eye disorders) | 0 | 1 | 0
VITREOUS HAEMORRHAGE (Eye disorders) | 2 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 2
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 1 | 0 | 0
ILEUS (Gastrointestinal disorders) | 0 | 1 | 0
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 1 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1 | 0
CHEST PAIN (General disorders) | 0 | 2 | 0
DEATH (General disorders) | 0 | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1 | 0
PYREXIA (General disorders) | 0 | 1 | 0
BILE DUCT STONE (Hepatobiliary disorders) | 0 | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1 | 0
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 1 | 0
ARTHRITIS BACTERIAL (Infections and infestations) | 0 | 0 | 1
BACTERIAL SEPSIS (Infections and infestations) | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 0 | 2
ENDOPHTHALMITIS (Infections and infestations) | 0 | 2 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 0
PAROTITIS (Infections and infestations) | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0
SEPSIS (Infections and infestations) | 1 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION PSEUDOMONAL (Infections and infestations) | 1 | 0 | 0
DRUG TOXICITY (Injury, poisoning and procedural complications) | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 2 | 1 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
INTRAOCULAR PRESSURE INCREASED (Investigations) | 0 | 2 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 1
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 | 0 | 0
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LUNG CARCINOMA CELL TYPE UNSPECIFIED STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
T-CELL PROLYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
AUTONOMIC NERVOUS SYSTEM IMBALANCE (Nervous system disorders) | 0 | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 2
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 0 | 1
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 4 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 0 | 1
TESTICULAR PAIN (Reproductive system and breast disorders) | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
AORTIC STENOSIS (Vascular disorders) | 0 | 0 | 1
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 0 | 1
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 1 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 0 | 1
LABILE HYPERTENSION (Vascular disorders) | 0 | 1 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (Sham) (N=189) | Ranibizumab (0.3 mg) (N=210) | Ranibizumab (0.5 mg) (N=203)
CATARACT (Eye disorders) | 4 | 11 | 11
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 29 | 37 | 31
CYSTOID MACULAR OEDEMA (Eye disorders) | 8 | 10 | 12
EYE PAIN (Eye disorders) | 12 | 7 | 12
MACULAR OEDEMA (Eye disorders) | 13 | 23 | 19
MACULOPATHY (Eye disorders) | 21 | 19 | 19
RETINAL DEPIGMENTATION (Eye disorders) | 11 | 13 | 4
RETINAL EXUDATES (Eye disorders) | 11 | 12 | 15
RETINAL HAEMORRHAGE (Eye disorders) | 33 | 54 | 51
RETINAL VASCULAR DISORDER (Eye disorders) | 19 | 29 | 21
VISUAL ACUITY REDUCED (Eye disorders) | 7 | 14 | 6
VITREOUS DETACHMENT (Eye disorders) | 9 | 9 | 15
BRONCHITIS (Infections and infestations) | 7 | 8 | 11
NASOPHARYNGITIS (Infections and infestations) | 14 | 13 | 8
SINUSITIS (Infections and infestations) | 8 | 11 | 9
URINARY TRACT INFECTION (Infections and infestations) | 7 | 12 | 10
INTRAOCULAR PRESSURE INCREASED (Investigations) | 9 | 15 | 12
HYPERTENSION (Vascular disorders) | 14 | 21 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No